CLINICAL TRIAL: NCT06096844
Title: A Randomized Phase III Trial of Chemo-Immunotherapy vs Immunotherapy Alone for the Vulnerable Older Adult With Advanced Non-Small Cell Lung Cancer: The ACHIEVE Study
Brief Title: Chemotherapy Combined With Immunotherapy Versus Immunotherapy Alone for Older Adults With Stage IIIB-IV Lung Cancer, The ACHIEVE Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-08628; NCI-2023-08628 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA5221 (Other: ECOG-ACRIN Cancer Research Group); EA5221 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2023-10-21; First posted 2023-10-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Advanced Lung Non-Small Cell Carcinoma; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — Carboplatin; Magnetic Resonance Spectroscopy; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes; Paclitaxel; pembrolizumab; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (pembrolizumab) (Active Comparator): INDUCTION: Patients receive pembrolizumab IV over 30 minutes on day 1 of each cycle. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients receive pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 or 42 days for 2 years in the absence of disease progression or unacceptable toxicity.
  Patients undergo MRI at baseline and CT and/or PET on the trial at baseline and throughout the trial.
  Interventions: Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Pembrolizumab; Procedure: Positron Emission Tomography; Other: Questionnaire Administration
- Arm B (pembrolizumab, chemotherapy) (Experimental): See Detailed Description
  Interventions: Drug: Carboplatin; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Nab-paclitaxel; Drug: Paclitaxel; Biological: Pembrolizumab; Drug: Pemetrexed; Procedure: Positron Emission Tomography; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm B (pembrolizumab, chemotherapy)
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; ABI007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; Naveruclif; Paclitaxel Albumin; paclitaxel albumin-stabilized nanoparticle formulation; Paclitaxel Nanoparticle Albumin-bound; Paclitaxel Protein-Bound; Protein-bound Paclitaxel
  Arms: Arm B (pembrolizumab, chemotherapy)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm B (pembrolizumab, chemotherapy)
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
Drug: Pemetrexed — Given IV
  Other Names: MTA; Multitargeted Antifolate; Pemfexy
  Arms: Arm B (pembrolizumab, chemotherapy)
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial compares the effect of adding chemotherapy to immunotherapy (pembrolizumab) versus immunotherapy alone in treating patients with stage IIIB-IV lung cancer. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving pembrolizumab and chemotherapy may help stabilize lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate whether there is an improvement in overall survival (OS) with chemotherapy combined with pembrolizumab compared to single agent pembrolizumab in this vulnerable older adult patient population.

SECONDARY OBJECTIVES:

I. To evaluate any difference in progression free survival (PFS) with chemotherapy combined with pembrolizumab as compared to single agent pembrolizumab.

II. To evaluate the difference in PFS rate at 3 months and at 6 months with chemotherapy combined with pembrolizumab as compared to single agent pembrolizumab.

III. To evaluate the difference in best objective response rate using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria to assess whether chemotherapy combined with pembrolizumab results in improved response rates compared to treatment with single agent pembrolizumab.

IV. To evaluate toxicity in those treated with chemotherapy combined with pembrolizumab compared to those treated with single agent pembrolizumab.

V. To evaluate patient reported quality of life (QOL) evaluations between treatment arms.

EXPLORATORY OBJECTIVES:

I. To compare safety and tolerability between treatment arms. II. To explore factors within the pre-treatment geriatric assessment (GA) as predictors of toxicity and outcomes. To describe changes between the intended chemotherapy treatment planned versus treatment given and referrals placed by treating provider based on GA results.

III. To evaluate the assessment of a novel, composite fPFS score using disease progression/functional impairment assessment as a potential correlate to OS in this vulnerable population.

IV. To evaluate the correlation of 3-months PFS with OS as a potential surrogate of OS benefit.

V. To evaluate the correlation of 6-months PFS with OS as a potential surrogate of OS benefit.

VI. To assess elective dose intensity of chemotherapy of patients who receive doublet chemotherapy versus single agent chemotherapy.

EXPLORATORY CORRELATIVE OBJECTIVE:

I. To relate gut microbe abundances to treatment outcomes, toxicity, and geriatric assessments.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A:

INDUCTION: Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 of each cycle. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 or 42 days for 2 years in the absence of disease progression or unacceptable toxicity.

ARM B:

INDUCTION: Patients receive pembrolizumab IV over 30 minutes on day 1 of each cycle. Patients also receive investigator's choice of a chemotherapy regimen: 1) Pemetrexed IV over 10 minutes + carboplatin IV over 30-60 minutes on day 1 of each cycle; 2) Nab-paclitaxel IV over 30 on days 1, 8, and 15 of each cycle + carboplatin IV over 30-60 minutes on day 1 of each cycle; 3) Paclitaxel IV over 1 hour on day 1, 8, and 15 of each cycle or over 3 hours on day 1 of each cycle + carboplatin IV over 30-60 minutes on day 1 of each cycle; 4) Nab-paclitaxel IV over 30 minutes on days 1, 8 and 15 of each cycle; 5) Paclitaxel IV over 3 hours on day 1 of each cycle or over 1 hour on days 1, 8, and 15 of each cycle; or 6) Pemetrexed IV over 10 minutes on day 1 of each cycle. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 or 42 days for 2 years in the absence of disease progression or unacceptable toxicity.

All patients undergo magnetic resonance imaging (MRI) at baseline and computed tomography (CT) and/or positron emission tomography (PET) on the trial at baseline and throughout the trial.

After completion of study treatment, patients are followed up every 3 months if < 2 years from randomization and every 6 months if 2-5 years from Step 1 registration.

ELIGIBILITY:
Inclusion Criteria:

* STEP 1 REGISTRATION
* Patient must be ≥ 70 years of age
* Patient must have histologically or cytologically confirmed non-small cell lung cancer (NSCLC) with PD-L1 Tumor Proportion Score (TPS) range of 1-49%
* Patient must have Stage IIIB, IIIC or IV disease and not be candidates for combined chemo-radiation. NOTE: Prior chemo-radiation therapy (RT) for stage III with recurrence is allowed
* Patient must have a tumor that is negative for EGFR mutation/ALK translocations or other actionable first line mutations in which patients would receive first-line oral tyrosine kinase inhibitors
* Patient must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 2
* Patient must agree not to father children while on study and for 6 months after the last dose of protocol treatment
* Patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible
* Absolute neutrophil count (ANC) ≥ 1,500/uL (obtained within 14 days prior to Step 1 registration)
* Platelets ≥ 75,000/uL (obtained within 14 days prior to Step 1 registration)
* Hemoglobin (Hgb) ≥ 8.0 g/dL (obtained within 14 days prior to Step 1 registration)
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (obtained within 14 days prior to Step 1 registration)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 3.0 × institutional ULN (obtained within 14 days prior to Step 1 registration)
* Creatinine clearance (CrCL) ≥ 45 mL/min (estimated using Cockcroft-Gault method with actual body weight or measured) (obtained within 14 days prior to Step 1 registration)
* Human immunodeficiency virus (HIV)-infected patients on effective antiretroviral therapy with undetectable viral load within 6 months of Step 1 registration are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have undetectable HCV viral
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patient must be English or Spanish speaking to be eligible for the QOL component of the study

  * NOTE: Sites cannot translate the associated GA or QOL forms
* Patient must not have symptomatic central nervous system disease (CNS) metastases. Patients with a clinical history of CNS metastases or cord compression are eligible if they have been definitively treated and are clinically stable for at least 14 days prior to Step 1 registration and off all steroids for at least 24 hours prior to Step 1 registration. Patients with asymptomatic CNS metastases are eligible
* Patient must not have had any prior cytotoxic chemotherapy regimen for metastatic disease. Chemotherapy given in the setting of adjuvant therapy or locally advanced disease is allowed as long as treatment was completed, and they have fully recovered from treatment related adverse events prior to Step 1 registration
* Patient must not have had any prior immunotherapy for metastatic disease. Immunotherapy given in the setting of adjuvant therapy or locally advanced disease is allowed as long as treatment was completed greater than 6 months prior to Step 1 registration
* Patient must not have a history of uncontrolled autoimmune conditions with the following exceptions, which are allowed: alopecia, vitiligo, rheumatoid arthritis, psoriasis/psoriatic arthritis, Hashimoto's thyroiditis, lupus, inflammatory bowel disease
* Patient must not be on immunosuppressive medication, including steroids (if doses exceed the equivalent of prednisone 10 mg daily). Short courses of steroids which are discontinued prior to randomization are acceptable. Patients on inhaled, intranasal and/or topical steroids are eligible
* Patient must have baseline imaging done assessing all measurable or non-measurable sites of disease within 45 days prior to Step 1 registration
* Investigator must declare their intended chemotherapy regimen should their patient be randomized to Arm B (doublet versus[vs] singlet)
* STEP 2 RANDOMIZATION
* Patient must have completed the baseline Geriatric Assessment (GA) after Step 1 registration and prior to Step 2 randomization

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From randomization to death from any cause, and patients who are alive at the time of final analysis will be censored at the last date of contact, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method, and Cox proportional hazards models will be used to estimate hazard ratios. Comparison of OS will use a logrank test stratified on the randomization stratification factors with a one-sided type I error rate of 0.025. Other comparisons of groups will be made using the log rank test and Cox modeling.

SECONDARY OUTCOMES:
Progression free survival (PFS) | From randomization to documented disease progression per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or death from any cause, whichever occurs first, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method, and Cox proportional hazards models will be used to estimate hazard ratios.
Six month PFS | From randomization to documented disease progression per RECIST 1.1 or death from any cause, whichever occurs first, assessed at 6 months
  Defined as the proportion of patients who remained alive and progression-free at 6 months. Will be estimated using the Kaplan-Meier method, and Cox proportional hazards models will be used to estimate hazard ratios.
Best objective response | Up to 5 years
  Will be evaluated via RECIST 1.1 criteria. Best objective response rate is defined as the proportion of patients with measurable disease at baseline achieved complete response (CR) or partial response (PR) as best response from the start of the treatment until disease progression/recurrence or start of non-protocol therapy. Patients who do not start treatment and patients who do not have any follow-up disease evaluation and do not meet RECIST criteria for clinical progression are coded as not evaluable. Patients who are not evaluable are included in the calculation of response rates (as non-responders).
Incidence of adverse events | Up to 2 years
  Toxicity will be determined using the Common Terminology Criteria for Adverse Events (CTCAE). Toxicity will be assessed by summaries by CTCAE grade.
Evaluation of quality of life (QOL) measures | Baseline up to 6 months
  Quality of life evaluations will be conducted using questionnaires at time of disease evaluation per Functional Assessment of Cancer Therapy-Lung version 4. QOL assessment will be gathered and the changes in QOL between the two treatment arms will be compared using Wilcoxon rank sum test. The comparison of changes in QOL using Wilcoxon rank sum test will also be done at 6 months given the high mortality rate in this population and the expectation that we may see differences in OS by that timepoint. Point estimates of all endpoints will be accompanied by the corresponding 95% confidence intervals. Point estimates of OS and the corresponding 95% confidence intervals by sex, race and ethnicity will be provided.

OTHER OUTCOMES:
Gut microbe abundances | Baseline and after 4 cycles of initial treatment (Cycles = 21 days)
  Will relate gut microbe abundances to treatment outcomes, toxicity, and geriatric assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Megan A Baumgart, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (314):
- United States (314):
  - Highlands Oncology Group - Fayetteville, Fayetteville, Arkansas
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - Highlands Oncology Group - Rogers, Rogers, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente Fresno Orchard Plaza, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente- Modesto MOB II, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-Oakland, Oakland, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Malcom Randall Veterans Administration Medical Center, Gainesville, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Moffitt Cancer Center at Wesley Chapel, Wesley Chapel, Florida
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - University of Illinois, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - Saint Catherine Hospital, Indianapolis, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - William E Kahlert Regional Cancer Center/Sinai Hospital, Westminster, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute at Boston Medical Center - Brighton, Brighton, Massachusetts
  - Dana-Farber Cancer Institute at Foxborough, Foxborough, Massachusetts
  - Dana Farber-Merrimack Valley, Methuen, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional, Milford, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at South Shore, South Weymouth, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - Briarcliff, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - The Dana-Farber Cancer Institute at Londonderry, Londonderry, New Hampshire
  - Jefferson Cherry Hill Hospital, Cherry Hill, New Jersey
  - Inspira Medical Center Mullica Hill, Mullica Hill, New Jersey
  - Penn Medicine Princeton Health, Plainsboro, New Jersey
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - Glens Falls Hospital, Glens Falls, New York
  - Upstate Cancer Center at Oswego, Oswego, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - SUNY Upstate Medical Center-Community Campus, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Upstate Cancer Center at Verona, Verona, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - Durham VA Medical Center, Durham, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Memorial Hospital, Marysville, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Ann B Barshinger Cancer Institute, Lancaster, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Reading Hospital McGlinn Cancer Institute at Phoenixville, Phoenixville, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Ralph H Johnson VA Medical Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - White River Junction Veteran Administration Medical Center, White River Junction, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - VCU Health Tappahannock Hospital, Tappahannock, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - ThedaCare Cancer Care - Berlin, Berlin, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercyhealth Hospital and Cancer Center - Janesville, Janesville, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ThedaCare Regional Medical Center - Neenah, Neenah, Wisconsin
  - ThedaCare Cancer Care - New London, New London, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - ThedaCare Cancer Care - Oshkosh, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - ThedaCare Cancer Care - Shawano, Shawano, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Sheboygan Physicians Group, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - ThedaCare Cancer Care - Waupaca, Waupaca, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
"NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page."
URL: https://grants.nih.gov/policy/sharing.htm